CLINICAL TRIAL: NCT06089681
Title: Comparison of Trunk Muscle Activity, Muscle Strength, Muscle Endurance Between Sprinters With and Without Hamstring Strain Injury History
Brief Title: Comparison of Trunk Muscle Performance Between Sprinters With and Without Hamstring Strain Injury History
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Other Study IDs: YM111052F
Record Dates: First submitted 2022-06-28; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-04

CONDITIONS: Hamstring Injury
Keywords: Hamstring Strain Injury; Trunk Muscle Performance; Hip Muscle Performance; Sprinter

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hamstring strain injury history group: Sprinters who have ≥ twice hamstring strain injury occurrence in the past year
- Control group: Sprinters who match gender, age, BMI, dominant side, training experience, training frequency, PB in 100m with HSI history group and without any hamstring strain injury occurrence in the past year

SUMMARY:
The aim of this study is to:

1. Compare trunk muscle performance between sprinters with and without HSI history
2. Investigate whether running speed influences the differences on trunk muscle activity between these two groups

DETAILED DESCRIPTION:
Hamstring strain injury is one of the most common injuries in the lower extremities. As running speed increases, the force and load on the hamstring muscles significantly increase, thereby increasing the risk of injury. Trunk muscles are connected thigh muscles through the pelvis, and poor trunk muscle capacity of maintaining stability affect the muscle length of the lower limbs during movement, reducing their contractile tension and increasing the risk of injury. Earlier literature also indicated that poor trunk muscle performance is related to the occurrence of lower extremity sport injuries. However, literature on the relationship between trunk muscle performance and hamstring strain injury is scarce. Testing methods of existing research have failed to fully reflect the actual circumstances of sprinting. Moreover, previous studies have predominantly focused on soccer players. However, the running mechanics of soccer player and sprinter are slightly different. Currently, there is lack of research investigate the relationship between trunk muscle performance and hamstring strain injury in sprinters.Therefore, the aim of this study is to: (1) Compare trunk muscle performance between sprinters with and without HSI history, (2) nvestigate whether running speed influences the differences on trunk muscle activity between these two groups

ELIGIBILITY:
Inclusion Criteria of HSI history group:

* Have ≥ twice hamstring strain injury occurrence in the past year

Inclusion Criteria of control group:

* Without any hamstring strain injury occurrence in the past year
* Match gender, age, BMI, dominant side, training experience, training frequency, Personal best record in 100m with HSI history group

Exclusion Criteria of all subjects:

* Neurological, cardiorespiratory or systemic disorder
* Have low back pain history in the past year
* Scoliosis
* Sacroiliac joint dysfunction
* Complaints of pain on trunk & lower extremity
* Leg length difference > 2cm
* History of lower extremity surgery

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Age between 16 to 30 years old
  * Sprinters who specialize in 100, 200, 400 meters, or 100, 400 metres hurdles
  * Participates in sprint training ≥ three times a week
  * Without any pain when participation in sporting activity
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Surface electromyography (Noraxon TeleMyo sEMG System, Noraxon USA Inc, Scottdale, Ariz) | Immediately during the experiment
  Muscle activation of external oblique, internal oblique, erect spinae, gluteus maximus when sprinting on the treadmill at 40% and 60% maximal speeds
Isometric trunk flexor muscle strength (Pro 4, Biodex Medical Systems, Inc., Shirley, NY, United States) | Immediately during the experiment
  Isometric muscle strength of trunk flexor is measured with Biodex System 4 Pro™ in sitting position
Isometric trunk extensor muscle strength (Pro 4, Biodex Medical Systems, Inc., Shirley, NY, United States) | Immediately during the experiment
  Isometric muscle strength of trunk extensor is measured with Biodex System 4 Pro™ in sitting position
Isometric trunk rotator muscle strength (microFET®2 Digital Handheld Dynamometer) | Immediately during the experiment
  Isometric muscle strength of trunk rotator is measured with microFET in hook-lying position
Trunk flexor muscle endurance | Immediately during the experiment
  Muscle endurance of trunk flexor is measured with trunk muscle endurance test. It requires subjects to sit on the test bench and place the upper body against a support with an angle of 60˚ from the test bed. Both the knees and hips are flexed to 90˚. The arms are folded across the chest with hands placed on the opposite shoulder and toes are placed under toe straps. Subjects will be instructed to maintain the body position while the supporting wedge is pulled back 10cm to begin the test. The test ends when the upper body falls below the 60˚ angle. The time the subjects maintain will be recorded.
Trunk extensor muscle endurance | Immediately during the experiment
  Muscle endurance of trunk extensor is measured with Biering-Sorensen test. It requires subjects to lay prone with the lower body fixed to the test bed at the ankles, knees, and hips and the upper body extended in a cantelevered fashion over the edge of the test bench. The test bench surface is approximately 25cm above the surface of the floor. Subjects rest their upper bodies on the floor before the exertion. At the beginning of the exertion the upper limbs are held across the chest with the hands resting on the opposite shoulders, and the upper body is lifted off the floor until the upper torso is horizontal to the floor. Subjects are instructed to maintain the horizontal position as long as possible. The time the subjects maintain will be recorded.
Trunk lateral flexor muscle endurance | Immediately during the experiment
  Muscle endurance of trunk lateral flexor is measured with side bridge test. It requires subjects to lay on an exercise mat (thickness, 2.5cm) on their sides with legs extended. The top foot is placed in front of the lower foot on the mat for support. Subjects are instructed to support themselves lifting their hips off the mat to maintain a straight line over their full body length, and support themselves on one elbow and their feet. The uninvolved arm is held across the chest with hand placed on the opposite shoulder. The test ends when the hips returns to the exercise mat. The time the subjects maintain will be recorded.

OTHER OUTCOMES:
Isokinetic lower extremity muscle strength ratio (Pro 4, Biodex Medical Systems, Inc., Shirley, NY, United States) | Immediately during the experiment
  Muscle strength ratios of hamstrings eccentric contraction at 30 ˚/s angular velocity and quadriceps concentric contraction at 240 ˚/s angular velocity, quadriceps concentric contraction at 240 ˚/s angular velocity and hamstrings concentric contraction at 240 ˚/s angular velocity, bilateral hamstrings concentric contraction at 60 ˚/s angular velocity are measured
Hamstring flexibility | Immediately during the experiment
  Hamstring flexibility is measured with 90-90 active straight leg test. It requires subjects to lay on the bed with hip and knee 90 degrees flexion. Subjects are instructed to extend their knee with hip 90 degrees flexion as possible. The knee angle is measured as hamstring flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Beitou, Taiwan